CLINICAL TRIAL: NCT06438445
Title: Effects of Royal Jelly Supplementation on Inflammation and Cellular Senescence in Chronic Kidney Disease Patients Under Hemodialysis
Brief Title: Effects of Royal Jelly Supplementation in Chronic Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Interventional
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Kidney Failure, Chronic; Oxidative Stress; Hemodialysis
Keywords: Cellular Senescence; Renal Dialysis; Renal Insufficiency, Chronic; Oxidative Stress
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Jelly Group (Experimental): Patients with chronic kidney disease on hemodialysis will receive capsules containing 500mg of royal jelly/day for two months.
  Interventions: Dietary Supplement: Real Jelly
- Placebo group (Placebo Comparator): Patients with chronic kidney disease on hemodialysis will receive capsules containing 500mg of placebo/ day for two months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Real Jelly — Participants will receive 500mg of royal jelly capsules per day for two months.
  Arms: Real Jelly Group
Dietary Supplement: Placebo — Participants will receive 500mg of placebo capsules per day for two months.
  Arms: Placebo group

SUMMARY:
The objective of this study is to evaluate the effects of royal jelly on inflammation and cellular senescence in patients with chronic kidney disease (CKD) on hemodialysis (HD).

DETAILED DESCRIPTION:
Royal jelly is a substance produced in the hypopharyngeal glands of bees that operate young, and rich in bioactive compounds such as polyphenols, free fatty acids and exclusive peptides capable of mitigating inflammation and premature aging (genomic instability, mitochondrial dysfunction, shortening of telomeres) existing in patients with chronic kidney disease (CKD) on hemodialysis. However, to date there are no studies evaluating the effects of royal jelly on such complications in patients with RDC. Objectives: To evaluate the effects of royal jelly on inflammation and cellular senescence in patients with CKD. Methods: Clinical, longitudinal, randomized study, with washout and crossover period. Patients with CKD on HD received 140 mL bottles containing propolis and turmeric, and were instructed to take 10 mL/day (dosing cup), containing a dose equivalent to 110 mg/day of standardized green propolis extract (EPP-AF) plus 130 mg of curcuminoids/day or placebo for 8 weeks. After this supplementation, patients will enter the washout period (8 weeks) and after this period, the intervention group will receive placebo and vice versa. The collection of biological material (blood and feces) will be done before and after each study period. The mRNA expression of the transcription factors Nrf2 and NF-κB, as well as their target genes, antioxidant enzymes, inflammatory cytokines and the expression of genes and proteins that modulate the protein will be evaluated using rtPCR, western blotting and assay methods. multiplex. Uremic toxins from the intestinal microbiota such as indoxyl sulfate (IS), p-cresyl sulfate (p-CS) and Indole-3-acetic acid (IAA) will be confirmed by HPLC and plasma lipopolysaccharide (LPS) levels will be analyzed by ELISA. The determination of antioxidant capacity will be determined by the FRAP, ORAC AND DPPH methods. The analysis of the composition of the intestinal microbiota will be evaluated by high-throughput sequencing of the V4-V5 region of the 16S ribosomal RNA gene. Nutritional status and dietary intake will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients with CKD undergoing hemodialysis for more than 6 months
* patients with arteriovenous fistula (AVF) as vascular access.

Exclusion Criteria:

* pregnant,
* lactating,
* smoker
* patients using antibiotics and antioxidant supplements in the last three months
* patients with autoimmune and infectious diseases,
* patients with cancer, liver disease, and AIDS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Change in inflammatory biomarkers | 6 weeks
  Changes in the mRNA levels of Nrf2, Keap1, Bach1, NLPR3, NF-kB, HO-1, NQO1, p14, p16, p21 and p53 as well as VCAM, ICAM and E-selectin and TLR-4, TNFR and AhR receptors, which will be evaluated from peripheral blood mononuclear cells.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, Study Director — Universidade Federal Fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil